CLINICAL TRIAL: NCT01248832
Title: Smokers' Quitline for Asian Language Speakers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Shu-Hong Zhu, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R01CA104573-5; R01CA104573 (NIH)
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Smoking Cessation
Keywords: tobacco cessation; smoking cessation; telephone; self-help; smoking abstinence; tobacco use disorder; disparity
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Cessation; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telephone Counseling (Experimental): Telephone Counseling
  Interventions: Behavioral: Telephone Counseling; Behavioral: Self-Help Materials
- Self-help Materials (Active Comparator): Self-help Materials
  Interventions: Behavioral: Self-Help Materials

INTERVENTIONS:
Behavioral: Telephone Counseling — Counseling is conducted in Mandarin, Cantonese, Korean, or Vietnamese by counselors at the Helpline. The protocol used is similar to that proved efficacious. However, to make the counseling culturally appropriate for Asian language speakers, we: capitalizing on first contact, present the Helpline as a credible quit smoking program staffed by "experts", avoid the term "counseling" since it is associated with mental illness, and assume a more authoritative role and directive counseling style. Counseling is proactive (1st call is made by smoker, then subsequent calls are made by the counselor) to help reduce attrition. Counseling includes a 30-40 minute comprehensive pre-quit session plus up to 5 shorter follow-up calls (about 10 minutes) scheduled according to the probability of relapse.
  Arms: Telephone Counseling
Behavioral: Self-Help Materials — All subjects (both in the telephone counseling group and the materials-only group) receive self-help materials in teh appropriate language. Materials were created in-house, are written in the appropriate language, and cover the essentials of the quitting process such as motivation, physiological and emotional responses to quitting, nicotine in the body, quitting aids, quitting strategies (including those that might be culturally specific such as acupuncture or herbs), setting a quit date, planning, relapse prevention, differentiating between slips and relapse, long-term maintenance, and developing the nonsmoker self-image.

SUMMARY:
The study tested the effects of telephone counseling for smokers from three Asian language speaking groups: Chinese, Korean, and Vietnamese. The specific aims were to: 1) test the efficacy of a culturally appropriate counseling protocol for smokers calling the California Smokers' Helpline on the Chinese, Korean and Vietnamese lines, 2) examine whether intervention effects varied by cognitive and behavioral predictors of cessation success, 4) examine whether family involvement plays a role in quitting success, and 5) assess differences in counseling effect across the three ethnic groups.

DETAILED DESCRIPTION:
Asian Americans are among the least studied groups in smoking research, which has created a knowledge gap in understanding their behavior and in developing methods to help them quit. No efficacy data have been reported for telephone counseling of smokers who prefer to use Asian languages, although telephone intervention holds promise for these groups because of its convenience and its potential to reach large numbers of smokers. In this two-arm design subjects are stratified by language (Chinese, Korean, and Vietnamese) and randomized to telephone counseling (plus materials) or self-help materials only, which serves as the control. The study is significant in several ways. First, it provides timely information on a cessation approach for a traditionally under-served population (Asian language speakers). Second, effective telephone counseling can be widely applied because of the proliferation of quitlines with centralized services in recent years. Third, by targeting Asian language speakers this study addresses the issue of ethnic disparities, which has been identified by many (including the NCI Bypass Budget) as a research priority.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old,
* daily smoker,
* ready to quit within one month,
* first time caller,
* valid phone number,
* valid address,
* California (CA) resident,
* gave consent to participate in study and evaluation,
* called the Chinese, Korean or Vietnamese line

Exclusion Criteria:

* used other form of tobacco,
* major medical or psychiatric complication (e.g. lung cancer, major depressive disorder, anti-psychotic medicine, recent stroke, impending surgery)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2277 (Actual)
Dates: Start 2004-08; Primary Completion 2008-04 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Number of participants who are continuously abstinent from cigarettes | 7-months post enrollment
  Continuous abstinence from cigarettes

SECONDARY OUTCOMES:
Number of participants who are continuously abstinent from cigarettes | 4-months post enrollment
  Continuous abstinence from cigarettes
Rate of serious quit attempts | 4-months post enrollment
  Quit Attempts
30-day point prevalence | 4-months post enrollment
  30-day point prevalence
30-day point prevalence | 7-months post enrollment
  30-day point prevalence
Rate of serious quit attempts | 7-months post enrollment
  Quit Attempts

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Hong Zhu, Ph.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

REFERENCES:
- [Background] Zhu SH, Wong S, Stevens C, Nakashima D, Gamst A. Use of a smokers' quitline by Asian language speakers: results from 15 years of operation in California. Am J Public Health. 2010 May;100(5):846-52. doi: 10.2105/AJPH.2009.168385. Epub 2010 Mar 18. PMID 20299658